CLINICAL TRIAL: NCT04127331
Title: Ultrasonographic Evaluation of Gastric Volume and Contents Before Surgery in Children
Brief Title: Gastric Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alok Moharir (Other)
Responsible Party: Sponsor-Investigator, Alok Moharir, Clinical Assistant Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000480
Record Dates: First submitted 2019-10-14; First posted 2019-10-15 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-02

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine (Active Comparator): Patients who are scheduled for routine outpatient surgery.
  Interventions: Device: Point-of-Care Ultrasound
- Urgent (Active Comparator): Patients who are scheduled for urgent surgery.
  Interventions: Device: Point-of-Care Ultrasound
- Emergent (Active Comparator): Patients who are scheduled for emergency surgery.
  Interventions: Device: Point-of-Care Ultrasound

INTERVENTIONS:
Device: Point-of-Care Ultrasound — Portable ultrasonography done at the bedside.

SUMMARY:
The primary objective of this study is to evaluate gastric volume and contents as well as gall bladder size in patients scheduled for routine, urgent, and emergency surgery. The hypothesis is that patients with stress, pain and opioid administration will have delayed gastric emptying and therefore a larger gastric fluid volume than those scheduled for elective surgery. The patients who have an appropriate NPO time will have a larger gallbladder size than the patients with shorter NPO time.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients aged 2-18 years of scheduled for elective, urgent, or emergent surgery under general anesthesia.

Exclusion Criteria:

* History of upper gastro-intestinal surgery.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Elective: Patients who are scheduled for routine outpatient surgery.
  Point-of-Care Ultrasound: Portable ultrasonography done at the bedside.
- Semi-urgent: Patients who are scheduled for semi-urgent surgery - within 6 hours of admission.
  Point-of-Care Ultrasound: Portable ultrasonography done at the bedside.
- Urgent: Patients who are scheduled for urgent surgery - within 2 hours of admission.
  Point-of-Care Ultrasound: Portable ultrasonography done at the bedside.
Period: Overall Study
Arm/Group | Elective | Semi-urgent | Urgent
Started | 41 | 32 | 27
Completed | 41 | 32 | 27
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elective | Semi-urgent | Urgent | Total
Number analyzed (Participants) | 41 | 32 | 27 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41 | 32 | 27 | 100
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (5.3) | 9.8 (4.1) | 10.6 (3.1) | 9.2 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 11 | 40
  Male | 24 | 20 | 16 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 32 | 27 | 100
Weight [Mean (Standard Deviation); unit: kilograms] | 35.5 (16.8) | 44.1 (8) | 47.6 (17.5) | 41.5 (18)
BMI [Mean (Standard Deviation); unit: kg/m2] | 19.3 (4.1) | 21.3 (4.2) | 20.8 (4) | 20.3 (4.2)
American Society of Anesthesiologists (ASA) status [Median (Inter-Quartile Range); unit: units on a scale] — ASA I = Normal healthy patient, ASA II - Patient with mild systemic disease
  units on a scale | 2 [1 to 2] | 1 [1 to 2] | 2 [1 to 2] | 2 [1 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Aspiration Risk Grade
Description: Grade 0: No fluid visible in the gastric antrum Grade 1: Clear fluid visualized with volume < 1.5 mL/kg Grade 2: Clear fluid visualized with volume > 1.5 mL/kg (High risk of aspiration)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Elective | Semi-urgent | Urgent
Number analyzed (Participants) | 41 | 32 | 27
Participants
  0 | 30 | 30 | 20
  1 | 9 | 2 | 6
  Solid (High risk) | 1 | 0 | 0
  Inconclusive | 1 | 0 | 1

2. Secondary Outcome: NPO at the Time of Injury
Description: Amount of time the patient was without food or water prior to their injury. This only applies to the Semi-urgent and Urgent groups.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Semi-urgent | Urgent
Number analyzed (Participants) | 6 | 28
Participants
  < 8 hours | 1 | 6
  > 8 hours | 5 | 22

3. Secondary Outcome: NPO at the Time of Surgery
Description: Amount of time the patient was without food or water prior to their surgery.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Elective | Semi-urgent | Urgent
Number analyzed (Participants) | 41 | 32 | 27
Participants
  < 8 hours | 2 | 1 | 2
  > 8 hours | 39 | 31 | 25

4. Secondary Outcome: Pre-operative Opioid Administration
Description: Patients who received opioids for pain control prior to surgery.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Urgent: Patients who are scheduled for urgent surgery - within 1 hour of admission.
  Point-of-Care Ultrasound: Portable ultrasonography done at the bedside.
Arm/Group | Elective | Semi-urgent | Urgent
Number analyzed (Participants) | 41 | 32 | 27
Participants | 0 | 5 | 11

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Elective | Semi-urgent | Urgent
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/32 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/32 | 0/27
Other Adverse Events (participants affected / at risk) | 0/41 | 0/32 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT04127331/Prot_SAP_000.pdf